CLINICAL TRIAL: NCT03253744
Title: Phase I Trial of Image Guided Focally Dose Escalated Prostate SBRT for Locally Recurrent Prostate Cancer After Prior Radiotherapy
Brief Title: Prostate SBRT for Locally Recurrent Prostate Cancer After Prior Radiotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Citrin, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170153; 17-C-0153
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Prostatic Neoplasm
Keywords: Image Guidance; Dose Escalation; Radiotherapy; Re-irradiation; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; 18F-JK-PSMA-7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1, Level 1, Arm 1: Tumor Irradiation (Experimental): Arm 1: Tumor irradiation.
  Cohort 1, Level 1, Arm 1 - 40 gray (Gy) to Tumor planning target volume (PTV)
  Stereotactic body radiation therapy (SBRT) will be delivered to areas of recurrent prostate cancer identified on imaging and biopsy.
  External beam radiation therapy (EBRT): Participants with locally recurrent prostate cancer after treatment with EBRT. These participants cannot have had permanent brachytherapy as part of their treatment.
  Interventions: Drug: 18F-DCFPyL; Radiation: Tumor Irradiation
- Cohort 1, Level 2, Arm 1 - Tumor Irradiation (Experimental): Arm 1: Tumor irradiation.
  Cohort 1, Level 2, Arm 1 - 42.5 gray (Gy) to Tumor planning target volume (PTV)
  Stereotactic body radiation therapy (SBRT) will be delivered to areas of recurrent prostate cancer identified on imaging and biopsy; and a reduced dose will be delivered to the entire prostate.
  External beam radiation therapy (EBRT): Participants with locally recurrent prostate cancer after treatment with EBRT. These participants cannot have had permanent brachytherapy as part of their treatment.
  Interventions: Drug: 18F-DCFPyL; Radiation: Tumor Irradiation
- Cohort 2, Level 1, Arm 2 - Prostate and Tumor Irradiation (Experimental): Arm 2: Prostate and tumor irradiation
  Cohort 2, Level 1, Arm 2 - 30 gray (Gy) PTV to Prostate and 40 Gy to Tumor planning target volume (PTV)
  Stereotactic body radiation therapy (SBRT) will be delivered to areas of recurrent prostate cancer identified on imaging and biopsy; and a reduced dose will be delivered to the entire prostate.
  Brachytherapy: Participants with locally recurrent prostate cancer after treatment with brachytherapy +/- external beam radiation therapy (EBRT). These participants must have had brachytherapy as part of their treatment.
  Interventions: Drug: 18F-DCFPyL; Radiation: Prostate + tumor irradiation; Radiation: Tumor Irradiation
- Cohort 2, Level 2, Arm 2 - Prostate and Tumor Irradiation (Experimental): Arm 2: Prostate and tumor irradiation
  Arm 2 - 30 gray (Gy) planning target volume (PTV) to Prostate and 42.5 Gy to Tumor PTV
  Stereotactic body radiation therapy (SBRT) will be delivered to areas of recurrent prostate cancer identified on imaging and biopsy; and a reduced dose will be delivered to the entire prostate.
  Brachytherapy: Participants with locally recurrent prostate cancer after treatment with brachytherapy +/- external beam radiation therapy (EBRT). These participants must have had brachytherapy as part of their treatment.
  Interventions: Drug: 18F-DCFPyL; Radiation: Prostate + tumor irradiation; Radiation: Tumor Irradiation

INTERVENTIONS:
Drug: 18F-DCFPyL — Participants will receive 2-(3-{1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-amino]-pentyl}-ureido)-pentanedioic acid at baseline and 6 months after radiation. The maximum amount of injected active drug will be less than 4.02 micrograms. The target administered activity will be 6-6.5 mCi.
  Other Names: 2-(3-{1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-amino]-pentyl}-ureido)-pentanedioic acid
Radiation: Tumor Irradiation — Stereotactic body radiation therapy (SBRT) will be delivered to areas of recurrent prostate cancer identified on imaging and biopsy.
  Other Names: SBRT
  Arms: Cohort 1, Level 1, Arm 1: Tumor Irradiation; Cohort 1, Level 2, Arm 1 - Tumor Irradiation
Radiation: Prostate + tumor irradiation — Stereotactic body radiation therapy (SBRT) will be delivered to areas of recurrent prostate cancer identified on imaging and biopsy; and a reduced dose will be delivered to the entire prostate.
  Other Names: SBRT
  Arms: Cohort 2, Level 1, Arm 2 - Prostate and Tumor Irradiation; Cohort 2, Level 2, Arm 2 - Prostate and Tumor Irradiation
Radiation: Tumor Irradiation — External beam radiation therapy (EBRT): Participants with locally recurrent prostate cancer after treatment with EBRT. These participants cannot have had permanent brachytherapy as part of their treatment.
  Other Names: EBRT

SUMMARY:
Background:

Prostate cancer is the second leading cause of cancer death in United States (U.S.) men. Radiation is an effective treatment for most patients with localized prostate cancer, but sometimes the tumor returns. Researchers want to see if a highly focused type of radiation can help. It is given in only 5 treatments. It is called stereotactic body radiation therapy (SBRT).

Objective:

To study the maximum tolerated dose and side effects of stereotactic body radiation therapy in people with a local recurrence of prostate cancer after radiation.

Eligibility:

Men at least 18 years old who have recurrent prostate cancer after radiation therapy and no evidence of distant metastatic disease.

Design:

Participants will be screened with blood tests, physical exam, and medical history. They may also have:

Magnetic resonance imaging (MRI) scan of the prostate.

Positron emission tomography (PET)/computed tomography (CT) scan. Participants will get an injection of 2-(3-{1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-amino]-pentyl}-ureido)-pentanedioic acid (18F-DCFPyL) for the PET scan. They will lie very still on their back on the scanner table.

Small samples of prostate tumor tissue will be taken by a needle through the skin or rectum to see if the cancer is in the prostate. Small metal seeds will be placed into the prostate at the same time to help guide the radiation.

About 2 weeks later, participants will have a radiation treatment planning CT scan.

Participants will answer questions about their urine function, bowel function, erectile function, and mood.

Participants will receive SBRT. They will have 5 radiation treatments over 2 weeks.

Participants will have follow-up visits. They will have a physical exam, blood tests, and questionnaires.

Six months after ending SBRT, the 18F-DCFPyL PET/CT will be repeated.

Participants will continue to have routine visits until two years after treatment is completed....

DETAILED DESCRIPTION:
Background:

* Prostate cancer that recurs after prior radiation treatment can be challenging to cure due to the side effects of available treatments such as surgery and cryoablation.
* Re-irradiation with brachytherapy or stereotactic approaches has shown excellent rates of prostate cancer disease control with tolerable side effects.
* Using image guidance to allow highly conformal focal re-irradiation may potentially increase the efficacy of re-irradiation.

Objectives:

-Define the maximum tolerated dose (MTD) of image guided, focally dose escalated prostate radiation with stereotactic body radiation therapy (SBRT) in patients with a local recurrence of prostate cancer after prior radiotherapy.

Eligibility:

* Histological confirmation of recurrent prostate cancer after prior irradiation (external beam or brachytherapy)
* No evidence of distant metastases of prostate cancer
* No prior prostatectomy
* Subject is greater than or equal to18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).

Design:

* This is a Phase I trial of focal dose escalation with SBRT using image and pathologic guidance.
* Areas in the prostate shown to have tumor on biopsy or with advanced imaging studies will be treated with highly conformal SBRT over a period of two to three weeks. Treatment will be guided and gated by fiducials implanted in the prostate.
* Patients will be treated to escalating doses based on tolerability of the treatment.
* Quality of life and functional outcomes such as urine, bowel, and erectile function will be assessed with questionnaires.
* Up to 52 patients will be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed locally recurrent adenocarcinoma of the prostate after prior radiation (external beam radiation therapy (EBRT) or brachytherapy).
* Prostate-specific antigen (PSA) failure after definitive radiation as defined by the Phoenix criteria (PSA elevation at least 2 nanograms (ng) per deciliter (dL) above post-radiotherapy nadir)
* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* PSA greater than or equal to 20 ng/dL if no prior 2-(3-{1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-amino]-pentyl}-ureido)-pentanedioic acid (18F-DCFPyL) scan obtained (If PSA > 20 and 18F-DCFPyL obtained within 3 months prior to enrollment shows no evidence of metastatic disease, subjects may be included in the study)
* Biochemical recurrence within one year of completion of radiotherapy
* Need for chronic anticoagulation therapy (chronic low dose aspirin is not an exclusion)
* Pre-existing and ongoing radiation-related grade 3 bowel or bladder toxicity
* Inflammatory bowel disease
* Active Lupus or Active scleroderma
* Patients with distant metastatic disease (prostate adjacent adenopathy is not an exclusion)
* Prior prostatectomy
* Subjects with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results.
* Subjects with severe claustrophobia that is unresponsive to oral anxiolytics
* Other medical conditions deemed by the Principal Investigator (or associates) to make the subject unsafe or ineligible for protocol procedures
* Subjects weighing > 350 lbs. (weight limit for scanner table), or unable to fit within the imaging gantry
* Serum creatinine > 2 times the upper limit of normal
* Total bilirubin > 2 times the upper limit of normal OR in patients with Gilbert's syndrome, a total bilirubin > 3.0.
* Liver transaminases (alanine aminotransferase (ALT), aspartate aminotransferase (AST) greater than 3 times the upper limit of normal
* Patients with positive Human Immunodeficiency Virus (HIV) status and currently requiring treatment with agents known to sensitize to irradiation, such as protease inhibitors.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0153.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, Level 1, Arm 1: 40 Gray (Gy) Tumor Irradiation Prostate and Tumor: Arm 1: Tumor irradiation.
  Cohort 1, Level 1, Arm 1 - 40 gray (Gy) to Tumor planning target volume (PTV)
  External beam radiation therapy (EBRT): Participants with locally recurrent prostate cancer after treatment with EBRT. These participants cannot have had permanent brachytherapy as part of their treatment.
  All participants received stereotactic body radiation therapy (SBRT) and 2-(3-{ 1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-amino]-pentyl} -ureido)-pentanedioic acid.
- Cohort 1, Level 2, Arm 1 - 42.5 Gray (Gy) Tumor Irradiation: Arm 1: Tumor irradiation. Cohort 1, Level 2, Arm 1 - 42.5 gray (Gy) to Tumor planning target volume (PTV);
  External beam radiation therapy (EBRT): Participants with locally recurrent prostate cancer after treatment with EBRT. These participants cannot have had permanent brachytherapy as part of their treatment.
  All participants received stereotactic body radiation therapy (SBRT) and 2-(3-{ 1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-amino]-pentyl} -ureido)-pentanedioic acid.
- Cohort 2, Level 1, Arm 2 - 30 Gray (Gy) and 40 Gy Prostate and Tumor Irradiation: Arm 2: Prostate and tumor irradiation Cohort 2, Level 1, Arm 2 - 30 gray (Gy) planning target volume (PTV) to Prostate and 40Gy to Tumor PTV
  Brachytherapy: Participants with locally recurrent prostate cancer after treatment with brachytherapy +/- external beam radiation therapy (EBRT). These participants must have had brachytherapy as part of their treatment.
  All participants received stereotactic body radiation therapy (SBRT) and 2-(3-{ 1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-amino]-pentyl} -ureido)-pentanedioic acid.
- Cohort 2, Level 2, Arm 2 - 30 Gray (Gy) and 42.5 Gy Prostate and Tumor Irradiation: Arm 2: Prostate and tumor irradiation Arm 2 - 30 gray (Gy) planning target volume (PTV) to Prostate and 42.5 Gy to Tumor PTV
  Brachytherapy: Participants with locally recurrent prostate cancer after treatment with brachytherapy +/- external beam radiation therapy (EBRT). These participants must have had brachytherapy as part of their treatment.
  All participants received stereotactic body radiation therapy (SBRT) and 2-(3-{ 1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-amino]-pentyl} -ureido)-pentanedioic acid.
Period: SBRT Treatment
Arm/Group | Cohort 1, Level 1, Arm 1: 40 Gray (Gy) Tumor Irradiation Prostate and Tumor | Cohort 1, Level 2, Arm 1 - 42.5 Gray (Gy) Tumor Irradiation | Cohort 2, Level 1, Arm 2 - 30 Gray (Gy) and 40 Gy Prostate and Tumor Irradiation | Cohort 2, Level 2, Arm 2 - 30 Gray (Gy) and 42.5 Gy Prostate and Tumor Irradiation
Started | 6 | 2 | 3 | 6
Completed | 6 | 2 | 3 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Completed Dose-Limiting Toxicity Assess.
Arm/Group | Cohort 1, Level 1, Arm 1: 40 Gray (Gy) Tumor Irradiation Prostate and Tumor | Cohort 1, Level 2, Arm 1 - 42.5 Gray (Gy) Tumor Irradiation | Cohort 2, Level 1, Arm 2 - 30 Gray (Gy) and 40 Gy Prostate and Tumor Irradiation | Cohort 2, Level 2, Arm 2 - 30 Gray (Gy) and 42.5 Gy Prostate and Tumor Irradiation
Started | 6 | 2 | 3 | 6
Completed | 6 | 2 | 3 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Completion of Follow-Up
Arm/Group | Cohort 1, Level 1, Arm 1: 40 Gray (Gy) Tumor Irradiation Prostate and Tumor | Cohort 1, Level 2, Arm 1 - 42.5 Gray (Gy) Tumor Irradiation | Cohort 2, Level 1, Arm 2 - 30 Gray (Gy) and 40 Gy Prostate and Tumor Irradiation | Cohort 2, Level 2, Arm 2 - 30 Gray (Gy) and 42.5 Gy Prostate and Tumor Irradiation
Started | 6 | 2 | 3 | 6
Completed | 4 | 2 | 3 | 2
Not Completed | 2 | 0 | 0 | 4
Not completed — Continuing follow-up. | 2 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Level 1, Arm 1: 40 Gray (Gy) Tumor Irradiation Prostate and Tumor | Cohort 1, Level 2, Arm 1 - 42.5 Gray (Gy) Tumor Irradiation | Cohort 2, Level 1, Arm 2 - 30 Gray (Gy) and 40 Gy Prostate and Tumor Irradiation | Cohort 2, Level 2, Arm 2 - 30 Gray (Gy) and 42.5 Gy Prostate and Tumor Irradiation | Total
Number analyzed (Participants) | 6 | 2 | 3 | 6 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 2 | 3
  >=65 years | 5 | 2 | 3 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.02 (5.65) | 78.3 (5.66) | 72.7 (4.17) | 65.95 (4.51) | 70.38 (6.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 2 | 3 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 3 | 6 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 0 | 1 | 5
  White | 2 | 2 | 3 | 5 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 3 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD of image-guided, focally dose escalated prostate stereotactic body radiation therapy (SBRT) in participants with a local recurrence of prostate cancer after prior radiotherapy. The MTD is the dose level at which no more than 1 of up to 6 participants experience dose-limiting toxicity (DLT) during treatment and up to 3 weeks following completion of treatment, and the dose below that at which at least 2 (of .6) participants have DLT as a result of treatment. A DLT is a Grade 3 rectal, small bowel, or urinary toxicity that does not resolve to Grade 2 or less within 4 days, other Grade 3 in-field toxicities attributable to Stereotactic body radiation therapy (SBRT) that do not resolve to a Grade 2 or less within 4 days, and delays of more than one week in completing radiation treatment due to toxicity.
Time Frame: 3 weeks post-treatment
Measure: Number; unit: gray (Gy)
Groups:
- All Participants in Arm 1: All participants in Arm1: 40 Gy Tumor irradiation who received at least one dose of stereotactic body radiation therapy (SBRT) are considered evaluable for toxicity. Only participants who have completed SBRT and have their prostate-specific antigen (PSA) measured are considered evaluable for response.
- All Participants in Arm 2: All participants in Arm 2. 42.5 Gy Tumor and 30 Gy Prostate irradiation who received at least one dose of stereotactic body radiation therapy (SBRT) are considered evaluable for toxicity. Only participants who have completed SBRT and have their prostate-specific antigen (PSA) measured are considered evaluable for response.
Arm/Group | All Participants in Arm 1 | All Participants in Arm 2
Number analyzed (Participants) | 8 | 9
gray (Gy) | 40 | 42.5

2. Secondary Outcome: Sensitivity of 2-(3-{1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-Amino]-Pentyl}-Ureido)-Pentanedioic Acid (18F-DCFPyL) Imaging as Compared to Biopsy in Detecting Locally Recurrent Prostate Cancer
Description: The sensitivity of DCF-PyL for detecting locally recurrent prostate cancer (at baseline) will be reported using biopsy as the gold standard to evaluate 18F-DCFPyL imaging as a method to detect locally recurrent prostate cancer after radiation. Sensitivity is the number of true positives divided by the sum of the number of true positives and false negatives. Lesions detected on DCF-PyL that are biopsy confirmed are considered true positives. Lesions that are not detected on DCFPyL and are biopsy positive are considered false negatives.
Time Frame: 6 months after radiation
Measure: Number (95% Confidence Interval); unit: Percent
Groups:
- All Participants in Arm 1: All participants in Arm1 who received at least one dose of stereotactic body radiation therapy (SBRT) are considered evaluable for toxicity. Only participants who have completed SBRT and have their prostate-specific antigen (PSA) measured are considered evaluable for response.
- All Participants in Arm 2: All participants in Arm 2 who received at least one dose of stereotactic body radiation therapy (SBRT) are considered evaluable for toxicity. Only participants who have completed SBRT and have their prostate-specific antigen (PSA) measured are considered evaluable for response.
Arm/Group | All Participants in Arm 1 | All Participants in Arm 2
Number analyzed (Participants) | 8 | 9
Percent | 95 [82 to 99] | 100 [88 to 100]

3. Secondary Outcome: Specificity of 2-(3-{1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-Amino]-Pentyl}-Ureido)-Pentanedioic Acid (18F-DCFPyL) Imaging as Compared to Biopsy in Detecting Locally Recurrent Prostate Cancer
Description: The specificity of DCF-PyL for detecting locally recurrent prostate cancer (at baseline) will be reported using biopsy as the gold standard to evaluate 18F-DCFPyL imaging as a method to detect locally recurrent prostate cancer after radiation. Specificity is the number of true negatives divided by the sum of the number of true negatives and the number of false positives. Lesions that are not detected on DCF-PyL that are biopsy confirmed to have no tumor are considered true negatives. Lesions that are detected on DCF-PyL and are biopsy negative are considered false positives.
Time Frame: 6 months after radiation
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | All Participants in Arm 1 | All Participants in Arm 2
Number analyzed (Participants) | 8 | 9
Percent | 100 [96 to 100] | 100 [96 to 100]

4. Secondary Outcome: Changes of Sexual Health Inventory for Men (SHIM) Quality of Life (QOL) Scores During and After Treatment
Description: Changes of QOL scores during and after treatment of focally dose escalated prostate stereotactic body radiation therapy (SBRT) on participant reported outcomes (Sexual Health Inventory for Men (SHIM), in participants previously treated with radiotherapy. The QOL scores will be summarized at baseline and for each visit. Linear mixed effects model will be used to model quality of life scores at baseline and during and after treatment in which random intercept and random slope are used to account for participant-specific trajectory of QOL scores. The SHIM is a 5-question quiz used to identify erectile dysfunction and assess its severity. The composite score is generated by adding the score for each question. The total score can range from 1-25. Higer values represent better erectile function.
Time Frame: Baseline compared to 24 months after treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | All Participants in Arm 1 | All Participants in Arm 2
Number analyzed (Participants) | 8 | 9
Scores on a scale
  Baseline | 7.25 (8.36) | 14.33 (10.44)
  After treatment | 5.75 (7.61) | 6.71 (9.10)

5. Secondary Outcome: Changes of American Urologic Association (AUA) Symptom Index Quality of Life (QOL) Scores During and After Treatment
Description: Changes of QOL scores during and after treatment of focally dose escalated prostate stereotactic body radiation therapy (SBRT) on participant reported outcomes, American Urologic Association (AUA) Symptom Index, in participants previously treated with radiotherapy. The QOL scores will be summarized at baseline and for each visit. Linear mixed effects model will be used to model quality of life scores at baseline and during and after treatment in which random intercept and random slope are used to account for participant-specific trajectory of QOL scores. The AUA Symptom Index is a 7-question quiz used to identify urinary symptoms and assess severity. Each question is scored based on the frequency of a different urinary symptoms. The composite score is generated by adding the score for each question. The total score can range from 0-35. Lower values represent less symptoms.
Time Frame: Baseline compared to 24 months after treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- All Participants in Arm 1: All participants in Arm 1 who received at least one dose of stereotactic body radiation therapy (SBRT) are considered evaluable for toxicity. Only participants who have completed SBRT and have their prostate-specific antigen (PSA) measured are considered evaluable for response.
Arm/Group | All Participants in Arm 1 | All Participants in Arm 2
Number analyzed (Participants) | 3 | 6
Scores on a scale
  Baseline | 5.75 (5.48) | 8.77 (6.53)
  After treatment | 11.86 (9.56) | 8.14 (3.98)

6. Secondary Outcome: Changes of Expanded Prostate Cancer Index Composite (EPIC-26) Quality of Life (QOL) Scores During and After Treatment
Description: Changes of QOL scores during and after treatment on participant reported outcomes, EPIC-26 in participants previously treated with radiotherapy. The QOL scores will be summarized at baseline and for each visit. Linear mixed effects model will be used to model QOL scores at baseline and during and after treatment in which random intercept and random slope are used to account for participant-specific trajectory of QOL scores. The EPIC-26 is a shortened, validated questionnaire used to assess health related QOL in individuals with prostate cancer. The EPIC-26 measures sexual function, bowel function, hormone therapy side effects, urinary incontinence, and urinary irritative symptoms. The survey has 26 individual items that have 4 to 5 response options that reflect a range of function from poor to excellent. The EPIC-26 uses a Likert scale for each item, and scores are transformed to a 0-100 scale, with higher scores indicating better Health-Related Quality of Life.
Time Frame: Baseline compared to 24 months after treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | All Participants in Arm 1 | All Participants in Arm 2
Number analyzed (Participants) | 8 | 9
Scores on a scale
  Baseline | 93.75 (11.57) | 75.00 (25.00)
  After treatment | 82.14 (27.82) | 71.43 (22.49)

7. Secondary Outcome: Biochemical Progression Free Survival (bPFS)
Description: bPFS, prostate-specific antigen (PSA) < 2 ng/dL above post stereotactic body radiation therapy (SBRT) nadir) at 1 and 2 years after treatment with focally dose escalated SBRT for locally recurrent prostate cancer after irradiation: bPFS will be estimated by the Kaplan-Meier survival analysis and effects of clinical variables on bPFS will be assessed by the Cox proportional hazards model. bPFS is defined as the duration of time from start of treatment to time of PSA progression or death, whichever occurs first. PSA progression (also known as biochemical failure) is defined based on elevation of PSA 2 ng/dL beyond the post-treatment nadir PSA, using the Phoenix criteria.
Time Frame: 1 and 2 years after treatment
Measure: Number; unit: percentage of participants
Arm/Group | All Participants in Arm 1 | All Participants in Arm 2
Number analyzed (Participants) | 8 | 9
percentage of participants
  1 year after treatment | 100 | 100
  2 years after treatment | 87.5 | 100

8. Secondary Outcome: Dose Limiting Toxicities (DLT)
Description: DLT's of image-guided, focally dose escalated prostate Stereotactic body radiation therapy (SBRT) in participants previously treated with radiotherapy. A DLT (during treatment and within the first three weeks after treatment) is defined as a Grade 3 rectal, small bowel, or urinary toxicity that does not resolve to Grade 2 or less within 4 days with appropriate medical management. Other grade 3 in-field toxicities attributable to SBRT that do not resolve to Grade 2 or less within 4 days with appropriate medical management. Delays of more than one week in completing radiation treatment due to toxicity. Toxicities were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Grade 2 is moderate. Grade 3 is severe.
  Define the dose-limiting toxicities and toxicity profile of image-guided, focally dose escalated prostate SBRT in patients previously treated with radiotherapy: DLTs will be reported descriptively.
Time Frame: 3 weeks after end of treatment
Measure: Number; unit: toxicities
Arm/Group | All Participants in Arm 1 | All Participants in Arm 2
Number analyzed (Participants) | 8 | 9
toxicities
  Grade 3 Cystitis non-infective | 1 | 0
  Grade 3 Urinary incontinence | 1 | 0

9. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 38 months (mos) & 26 days (d) for Cohort 1, Level 1, Arm 1, 29 mos & 9 d for Cohort 1, Level 2, Arm 1, 43 mos & 12 d for Cohort 2, Level 1, Arm 1, & 26 mos & 9 d for Cohort 2, Level 2, Arm 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Level 1, Arm 1: 40 Gray (Gy) Tumor Irradiation Prostate and Tumor | Cohort 1, Level 2, Arm 1 - 42.5 Gray (Gy) Tumor Irradiation | Cohort 2, Level 1, Arm 2 - 30 Gray (Gy) and 40 Gy Prostate and Tumor Irradiation | Cohort 2, Level 2, Arm 2 - 30 Gray (Gy) and 42.5 Gy Prostate and Tumor Irradiation
Number analyzed (Participants) | 6 | 2 | 3 | 6
Participants | 6 | 2 | 3 | 6

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 38 months and 26 days for Cohort 1, Level 1, Arm 1, 29 months and 9 days for Cohort 1, Level 2, Arm 1, 43 months and 12 days for Cohort 2, Level 1, Arm 1, and 26 months and 9 days for Cohort 2, Level 2, Arm 1.
Groups:
- Cohort 2, Level 2, Arm 2 - 30 Gray (Gy) and 42.5 Gy Prostate and Tumor Irradiation: AArm 2: Prostate and tumor irradiation Arm 2 - 30 gray (Gy) planning target volume (PTV) to Prostate and 42.5 Gy to Tumor PTV
  Brachytherapy: Participants with locally recurrent prostate cancer after treatment with brachytherapy +/- external beam radiation therapy (EBRT). These participants must have had brachytherapy as part of their treatment.
  All participants received stereotactic body radiation therapy (SBRT) and 2-(3-{ 1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-amino]-pentyl} -ureido)-pentanedioic acid.
Arm/Group | Cohort 1, Level 1, Arm 1: 40 Gray (Gy) Tumor Irradiation Prostate and Tumor | Cohort 1, Level 2, Arm 1 - 42.5 Gray (Gy) Tumor Irradiation | Cohort 2, Level 1, Arm 2 - 30 Gray (Gy) and 40 Gy Prostate and Tumor Irradiation | Cohort 2, Level 2, Arm 2 - 30 Gray (Gy) and 42.5 Gy Prostate and Tumor Irradiation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/2 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Level 1, Arm 1: 40 Gray (Gy) Tumor Irradiation Prostate and Tumor (N=6) | Cohort 1, Level 2, Arm 1 - 42.5 Gray (Gy) Tumor Irradiation (N=2) | Cohort 2, Level 1, Arm 2 - 30 Gray (Gy) and 40 Gy Prostate and Tumor Irradiation (N=3) | Cohort 2, Level 2, Arm 2 - 30 Gray (Gy) and 42.5 Gy Prostate and Tumor Irradiation (N=6)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Level 1, Arm 1: 40 Gray (Gy) Tumor Irradiation Prostate and Tumor (N=6) | Cohort 1, Level 2, Arm 1 - 42.5 Gray (Gy) Tumor Irradiation (N=2) | Cohort 2, Level 1, Arm 2 - 30 Gray (Gy) and 40 Gy Prostate and Tumor Irradiation (N=3) | Cohort 2, Level 2, Arm 2 - 30 Gray (Gy) and 42.5 Gy Prostate and Tumor Irradiation (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, supraventricular ectopy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 2 (2) | 1 (3) | 1 (1) | 5 (11)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, Diplopia, intermittent (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (2) | 0 (0) | 4 (4)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (2) | 2 (3)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Prostatic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, slow urine flow (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, weak stream (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Reproductive system and breast disorders - Other, Penile and perineal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, Priapism (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, nodule/cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (3) | 1 (1) | 3 (4)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT03253744/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT03253744/ICF_001.pdf